CLINICAL TRIAL: NCT01234688
Title: Effects of Aerobic Training During Hemodialysis on Exercise Tolerance in End Stage Renal Disease Patients
Brief Title: Effects of Aerobic Training in End Stage Renal Disease Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Juiz de Fora (Other)
Responsible Party: Maycon de Moura Reboredo, DSc, Federal University of Juiz de Fora
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2010-11-03; First posted 2010-11-04 (Estimated); Last update posted 2010-11-04 (Estimated); Status verified 2010-07

CONDITIONS: Kidney Failure, Chronic
Keywords: Exercise Tolerance; Physical Endurance
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exercise training (Experimental): Patients included in the exercise group were submitted to intra-dialytic exercise training, 3 times per week for 12 weeks.
  Interventions: Other: Exercise training
- Control (No Intervention): Patients allocated to the control group remained in regular dialysis treatment during the same timeframe.

INTERVENTIONS:
Other: Exercise training — Patients included in the exercise group were submitted to intra-dialytic exercise training, 3 times per week for 12 weeks.
  Other Names: Exercise group
  Arms: Exercise training

SUMMARY:
The investigators raised the hypothesis that exercise training would be associated with improvement in exercise tolerance and VO2 kinetics in hemodialysis patients.

DETAILED DESCRIPTION:
End-stage renal disease (ESRD) is associated with several hemodynamic and peripheral muscle abnormalities which could slow the kinetics of O2 uptake(VO2)and diminished tolerance to incremental exercise. Although previous studies have shown that aerobic training is able to accelerate VO2 kinetics in several disease populations, little is known if these positive findings are also applicable to hemodialysis patients.

ELIGIBILITY:
Inclusion Criteria:

The sample included end stage renal disease patients undergoing hemodialysis, three times per week totaling 12h weekly, for at least 6 months in the Nephrology Unit at the University Hospital of the Federal University of Juiz de Fora, State of Minas Gerais, Brazil. No patient had been involved in any kind of exercise training in the preceding 6 months

Exclusion Criteria:

* unstable angina;
* uncontrolled arrhythmia;
* uncompensated heart failure;
* uncontrolled hypertension (systolic blood pressure ≥ 200 mmHg and/or diastolic blood pressure ≥ 120 mmHg);
* diabetes mellitus;
* severe respiratory diseases;
* acute infection;
* severe renal osteodystrophy;
* neurological or musculoskeletal disturbances

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2008-06; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Effects of aerobic training during hemodialysis on exercise tolerance and VO2 kinetics in end stage renal disease patients | 3 months
  Before and after the intervention or control periods, the participants were submitted to an incremental work rate test and, two days apart, to a constant work rate test to the limit of tolerance.

CONTACTS AND LOCATIONS:
Overall Officials: Maycon M Reboredo, DSc, Principal Investigator — Federal University of Juiz de Fora; Rogério B de Paula, DSc, Study Director — Federal University of Juiz de Fora
Locations (1):
- Federal University of Juiz de Fora-Núcleo Interdisciplinar de Estudos e Pesquisas em Nefrologia (NIEPEN), Juiz de Fora, Minas Gerais, Brazil

REFERENCES:
- [Derived] Bernier-Jean A, Beruni NA, Bondonno NP, Williams G, Teixeira-Pinto A, Craig JC, Wong G. Exercise training for adults undergoing maintenance dialysis. Cochrane Database Syst Rev. 2022 Jan 12;1(1):CD014653. doi: 10.1002/14651858.CD014653. PMID 35018639
- [Derived] Reboredo MM, Neder JA, Pinheiro BV, Henrique DM, Lovisi JC, Paula RB. Intra-dialytic training accelerates oxygen uptake kinetics in hemodialysis patients. Eur J Prev Cardiol. 2015 Jul;22(7):912-9. doi: 10.1177/2047487314543079. Epub 2014 Jul 18. PMID 25038079
- [Derived] Reboredo MM, Neder JA, Pinheiro BV, Henrique DM, Faria RS, Paula RB. Constant work-rate test to assess the effects of intradialytic aerobic training in mildly impaired patients with end-stage renal disease: a randomized controlled trial. Arch Phys Med Rehabil. 2011 Dec;92(12):2018-24. doi: 10.1016/j.apmr.2011.07.190. PMID 22133251